CLINICAL TRIAL: NCT00176735
Title: Pilot Trial of Capecitabine and Radiation Therapy With Pre and Post Combination Chemotherapy in Advanced Pancreatic Cancer
Brief Title: Capecitabine and Radiation Therapy in Advanced Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2001-046
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine

INTERVENTIONS:
Drug: Capecitabine

SUMMARY:
Pancreatic cancer has traditionally been treated with chemotherapy and radiation therapy with limited results. Preliminary studies of parts of this program in patients with advanced pancreatic cancer have produced favorable results with acceptable side effects. We feel that this treatment sequence may help to slow and/or control the growth of pancreatic cancer.

This study will help doctors learn whether pancreatic cancer will respond to this treatment. This study will use the combination of two chemotherapy drugs, gemcitabine and cisplatin, before and after treatment with radiation therapy and an oral chemotherapy drug called capecitabine. This sequence of combination chemotherapy before and after radiation therapy, and radiation therapy with the drug capecitabine is what is under study. Parts of this sequence, for example, the combination of gemcitabine and cisplatin, have shown promising results in the treatment of pancreatic cancer. This research study is an attempt to combine these various parts.

ELIGIBILITY:
Eligibility Criteria

1. Patients must have cytologic or histologic confirmation of pancreatic carcinoma.
2. Patients must have unresectable disease with or without distant metastases. A status of unresectable will be based on review of helical CT scan and surgical consultation.
3. Patients with a history of previous abdominal irradiation or chemotherapy for pancreatic cancer are ineligible.
4. Patients must have an estimated life expectancy of at least 12 weeks and a Zubrod performance status of ≤ 2 (appendix I).
5. Patients must be 18 years of age or older. Patients with reproductive potential must agree to use an effective contraceptive method during treatment.
6. Patients must have adequate organ function defined as follows: bone marrow - granulocytes ≥ 1500/cmm, platelets > 100,000/cmm, renal - serum Cre < 1.5 mg/dl, hepatic - bilirubin < 3 mg/dl.
7. Patients must be free of other active systemic malignancy or any other serious co-morbid medical or psychiatric condition that would interfere with safe delivery of protocol therapy.
8. Patients must be aware of the investigational nature of the therapy and provide written informed consent as per institutional guidelines prior to the initiation of treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2001-12; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, M.D., Principal Investigator — University of Michigan Rogel Cancer Center